CLINICAL TRIAL: NCT07045168
Title: Risk-adapted Therapeutic Strategy in +1q NDMM： a Prospective, Multicenter Study
Brief Title: Risk-adapted Therapeutic Strategy in +1q NDMM
Status: Not yet recruiting | Type: Observational
Sponsor: FengYan Jin (Other)
Responsible Party: Sponsor-Investigator, FengYan Jin, The First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: Risk-adapted therapy
Record Dates: First submitted 2025-06-18; First posted 2025-07-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Risk-adapted therapeutic strategy; +1q MM; high-risk MM; minimal residual disease
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood、bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- low-risk +1q NDMM patients: This system classifies +1q NDMM patients into low, intermediate, and high-risk groups based on coexisting International Staging System (ISS) stage III, hypercalcemia, high lactate dehydrogenase (LDH), and t(14;16).Patients with ISS stage III, elevated LDH, hypercalcemia, and t(14;16) were assigned scores of 1 point, 1 point, 2 points, and 3 points, respectively. According to the tertiles of their scores,the patients with +1q were classified into low- (0 point) .
  Interventions: Other: risk-scoring model
- intermediate/high-risk +1q NDMM patients: This system classifies +1q NDMM patients into low, intermediate, and high-risk groups based on coexisting ISS stage III, hypercalcemia, high LDH, and t(14;16).Patients with ISS stage III, elevated LDH, hypercalcemia, and t(14;16) were assigned scores of 1 point, 1 point, 2 points, and 3 points, respectively. According to the tertiles of their scores,the patients with +1q was classified into intermediate- (1-3 points) and high-risk (4-7 points) groups.
  Interventions: Other: risk-scoring model
- 1q negativity low-risk group: Patients with 1q negativity were included as the control group, and patients were stratified into the high-risk group and low-risk group according to the 2025 IMWG Risk Stratification.
- 1q negativity high-risk group: Patients with 1q negativity were included as the control group, and patients were stratified into the high-risk group and low-risk group according to the 2025 IMWG Risk Stratification.

INTERVENTIONS:
Other: risk-scoring model — This system classifies +1q NDMM patients into low, intermediate, and high-risk groups based on coexisting ISS stage III, hypercalcemia, high LDH, and t(14;16).Patients with ISS stage III, elevated LDH, hypercalcemia, and t(14;16) were assigned scores of 1 point, 1 point, 2 points, and 3 points, respectively. According to the tertiles of their scores,the patients with +1q were classified into low- (0 point),intermediate- (1-3 points), and high-risk (4-7 points) groups.
  Other Names: Proposed risk-scoring model for estimating the prognostic impact of 1q gain in patients with newly diagnosed multiple myeloma
  Groups: intermediate/high-risk +1q NDMM patients; low-risk +1q NDMM patients

SUMMARY:
This real-world, multicenter prospective clinical study is designed to apply our internationally developed prognostic scoring system to guide individualized therapy in +1q newly diagnosed multiple myeloma (NDMM), using minimal residual disease (MRD) status as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18, or >=65 and fit according to IMWG-FI.
* Newly diagnosed NDMM by 2014 IMWG criteria.
* Adequate organ function for systemic therapy.
* Signed informed consent.

Exclusion Criteria:

* Active infections requiring systemic treatment.
* Unstable angina, NYHA class III-IV heart failure, or uncontrolled arrhythmias.
* History of hematologic or solid tumors treated with chemo/radiotherapy within 5 years.
* Current malignancies requiring therapy.
* Refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed NDMM by 2014 IMWG criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2029-07-04 (Estimated)

PRIMARY OUTCOMES:
MRD negativity rate | through study completion, up to 2 years
  To compare MRD negativity rate between low/intermediate- and high-risk +1q NDMM patients undergoing risk-adapted individualized treatment.
sustained MRD negativity rate | through study completion, up to 2 years
  To compare sustained MRD negativity rate between low/intermediate- and high-risk +1q NDMM patients undergoing risk-adapted individualized treatment.
Progression-Free Survival (PFS) | through study completion, up to 2 years
  PFS were calculated from the enrollment to the first instance of disease progression, relapse, or death
Overall Survival (OS) | through study completion, up to 2 years
  OS were calculated from the time of enrollment to death or the last follow-up
objective response rate | through study completion, up to 2 years
  To assess the objective response rate (ORR) and depth of response based on 2016 IMWG criteria (sCR, CR, VGPR, PR).
Treatment related adverse event(TRAE) | through study completion, up to 2 years
  Toxicity and safety will be reported based on the adverse events, as graded by CTCAE V5 and determined by routine clinical assessments.

SECONDARY OUTCOMES:
differences between MRD-negative and MRD-positive patients | through study completion, up to 2 years
  Number of participants with distinct immunological (T-cell subsets by flow cytometry), inflammatory (CRP, IL-6 levels), genomic (mutational burden by NGS), and proteomic (LC-MS/MS) signatures in MRD-negative vs. MRD-positive patients.
elderly +1q NDMM patients | through study completion, up to 2 years
  Number of participants achieving MRD negativity (by next-generation sequencing [NGS] at 10^-5 sensitivity) and progression-free survival (PFS) at 24 months in elderly intermediate/high-risk +1q NDMM patients receiving MRD-tailored therapy.
The efficacy of 1q negativity patients | through study completion, up to 2 years
  Patients with 1q negativity were included as the control group. According to the 2025 IMWG Risk Stratification, patients were divided into the high-risk group and the low-risk group. It is recommended that patients in the high-risk group receive CD38 monoclonal antibody in combination with the KRD regimen, while patients in the low-risk group receive CD38 monoclonal antibody in combination with the VRD regimen. The efficacy of these patients were compared with those of patients stratified by 1q risk through objective response rate (ORR) and depth of response based on 2016 IMWG criteria (sCR, CR, VGPR, PR) .
The survival of 1q negativity patients | through study completion, up to 2 years
  Patients with 1q negativity were included as the control group. According to the 2025 IMWG Risk Stratification, patients were divided into the high-risk group and the low-risk group. It is recommended that patients in the high-risk group receive CD38 monoclonal antibody in combination with the KRD regimen, while patients in the low-risk group receive CD38 monoclonal antibody in combination with the VRD regimen. The survival of these patients were compared with those of patients stratified by 1q risk through PFS and OS

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van de Donk NWCJ, Pawlyn C, Yong KL. Multiple myeloma. Lancet. 2021 Jan 30;397(10272):410-427. doi: 10.1016/S0140-6736(21)00135-5. PMID 33516340
- [Background] Zamagni E, Barbato S, Cavo M. How I treat high-risk multiple myeloma. Blood. 2022 May 12;139(19):2889-2903. doi: 10.1182/blood.2020008733. PMID 34727187
- [Background] Kumar SK, Rajkumar SV. The multiple myelomas - current concepts in cytogenetic classification and therapy. Nat Rev Clin Oncol. 2018 Jul;15(7):409-421. doi: 10.1038/s41571-018-0018-y. PMID 29686421
- [Background] Sonneveld P, Avet-Loiseau H, Lonial S, Usmani S, Siegel D, Anderson KC, Chng WJ, Moreau P, Attal M, Kyle RA, Caers J, Hillengass J, San Miguel J, van de Donk NW, Einsele H, Blade J, Durie BG, Goldschmidt H, Mateos MV, Palumbo A, Orlowski R. Treatment of multiple myeloma with high-risk cytogenetics: a consensus of the International Myeloma Working Group. Blood. 2016 Jun 16;127(24):2955-62. doi: 10.1182/blood-2016-01-631200. Epub 2016 Mar 21. PMID 27002115
- [Background] Croft J, Ellis S, Sherborne AL, Sharp K, Price A, Jenner MW, Drayson MT, Owen RG, Chown S, Lindsay J, Karunanithi K, Hunter H, Gregory WM, Davies FE, Morgan GJ, Cook G, Atanesyan L, Savola S, Cairns DA, Jackson G, Houlston RS, Kaiser MF. Copy number evolution and its relationship with patient outcome-an analysis of 178 matched presentation-relapse tumor pairs from the Myeloma XI trial. Leukemia. 2021 Jul;35(7):2043-2053. doi: 10.1038/s41375-020-01096-y. Epub 2020 Dec 1. PMID 33262523
- [Background] Wu J, Lu AD, Zhang LP, Zuo YX, Jia YP. [Study of clinical outcome and prognosis in pediatric core binding factor-acute myeloid leukemia]. Zhonghua Xue Ye Xue Za Zhi. 2019 Jan 14;40(1):52-57. doi: 10.3760/cma.j.issn.0253-2727.2019.01.010. Chinese. PMID 30704229
- [Background] D'Agostino M, Cairns DA, Lahuerta JJ, Wester R, Bertsch U, Waage A, Zamagni E, Mateos MV, Dall'Olio D, van de Donk NWCJ, Jackson G, Rocchi S, Salwender H, Blade Creixenti J, van der Holt B, Castellani G, Bonello F, Capra A, Mai EK, Durig J, Gay F, Zweegman S, Cavo M, Kaiser MF, Goldschmidt H, Hernandez Rivas JM, Larocca A, Cook G, San-Miguel JF, Boccadoro M, Sonneveld P. Second Revision of the International Staging System (R2-ISS) for Overall Survival in Multiple Myeloma: A European Myeloma Network (EMN) Report Within the HARMONY Project. J Clin Oncol. 2022 Oct 10;40(29):3406-3418. doi: 10.1200/JCO.21.02614. Epub 2022 May 23. PMID 35605179
- [Background] Abdallah NH, Binder M, Rajkumar SV, Greipp PT, Kapoor P, Dispenzieri A, Gertz MA, Baughn LB, Lacy MQ, Hayman SR, Buadi FK, Dingli D, Go RS, Hwa YL, Fonder AL, Hobbs MA, Lin Y, Leung N, Kourelis T, Warsame R, Siddiqui MA, Kyle RA, Bergsagel PL, Fonseca R, Ketterling RP, Kumar SK. A simple additive staging system for newly diagnosed multiple myeloma. Blood Cancer J. 2022 Jan 31;12(1):21. doi: 10.1038/s41408-022-00611-x. PMID 35102148
- [Background] Walker BA, Mavrommatis K, Wardell CP, Ashby TC, Bauer M, Davies F, Rosenthal A, Wang H, Qu P, Hoering A, Samur M, Towfic F, Ortiz M, Flynt E, Yu Z, Yang Z, Rozelle D, Obenauer J, Trotter M, Auclair D, Keats J, Bolli N, Fulciniti M, Szalat R, Moreau P, Durie B, Stewart AK, Goldschmidt H, Raab MS, Einsele H, Sonneveld P, San Miguel J, Lonial S, Jackson GH, Anderson KC, Avet-Loiseau H, Munshi N, Thakurta A, Morgan G. A high-risk, Double-Hit, group of newly diagnosed myeloma identified by genomic analysis. Leukemia. 2019 Jan;33(1):159-170. doi: 10.1038/s41375-018-0196-8. Epub 2018 Jul 2. PMID 29967379
- [Background] Yang P, Chen H, Liang X, Xu W, Yu S, Huang W, Yi X, Guo Q, Tian M, Yue T, Li M, Zhang Y, Zhang M, Yan Y, Hu Z, Kumar SK, Zhou F, Dai Y, Jin F. Proposed risk-scoring model for estimating the prognostic impact of 1q gain in patients with newly diagnosed multiple myeloma. Am J Hematol. 2023 Feb;98(2):251-263. doi: 10.1002/ajh.26774. Epub 2022 Nov 8. PMID 36309982